CLINICAL TRIAL: NCT03970876
Title: A Single Center, Randomized, Double-Blind, Active-controlled, Single-Dose, Phase I/II, Non-Inferiority Study Comparing ATGC-100 and Botox for the Treatment of Moderate to Severe Glabellar Lines in Adult Subjects
Brief Title: Safety and Efficacy Study of ATGC-100 for the Treatment of Moderate to Severe Glabellar Lines in Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBA-PLN-001
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2019-04

CONDITIONS: Moderate to Severe Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATGC-100 (Phase I/II) (Experimental): ATGC-100 will be injected to 5 glabellar lines (Each 4U/0.1ml, Total 20U/0.5ml)
  Interventions: Biological: ATGC-100
- Botox® (Phase II) (Active Comparator): Botox® will be injected to 5 glabellar lines (Each 4U/0.1ml, Total 20U/0.5ml)
  Interventions: Biological: Botox®

INTERVENTIONS:
Biological: ATGC-100 — Clostridium Botulinum Type A
  Arms: ATGC-100 (Phase I/II)
Biological: Botox® — Clostridium Botulinum Type A
  Arms: Botox® (Phase II)

SUMMARY:
Phase I/II clinical trial will be integrated and conducted. In phase I clinical trial, subjects with moderate to severe glabellar lines at maximum frown are enrolled and safety is assessed after 12 weeks of administration of 20U of ATGC-100. In phase II clinical trial, subjects with moderate to severe glabellar lines at maximum frown are enrolled, and efficacy and safety are assessed by comparing with Botox (Allergan).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged between 19 to 65 years old
2. Subjects attaining ≥ grade 2 in the investigator's rating of the severity of glabellar line at maximum frown
3. Subjects who voluntarily signed the informed consent

Exclusion Criteria:

1. Subjects with general neuromuscular synaptic disorders
2. Presence or history of eyelid and/or ptosis
3. Subjects with noticeable facial asymmetry
4. Inability to substantially lessen glabellar frown lines even by physically spreading apart
5. Subjects who have administered the following drugs within 4 weeks prior to screening: Muscle relaxants, Anti-cholinergic agents, Benzodiazepine and similar drugs, Benzamide drugs, Tetracycline antibiotics, Lincomycin antibiotics, Aminoglycoside antibiotics
6. Subjects who are taking Anti-Coagulant and Anti-Platelet agent
7. Subjects who have taken Aspirin and NSAIDs within 7 days prior to administration of investigational drug
8. Subjects with skin disorders at the injection site
9. Subjects with previous treatment of Face Lifting, Permanent Implant, and/or Filler in glabellar region
10. Subjects with prior filler treatments which would have interfered with the evaluation of the efficacy of the study treatment
11. Any other planned facial aesthetic procedure in the glabellar area during the trial period
12. Previous treatment with botulinum toxin in the forehead within the last 5 months or any planned treatment during the study period
13. A history of drug or alcohol abuse
14. Condition including anxiety disorder, or any other significant psychiatric disorder (e.g. depression), in the investigator's opinion

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE Version 5.0 (Phase I) | Up tp 12 weeks
Glabellar line improvement rate at maximum frown confirmed with investigator's assessment (Phase II) | 4 weeks after the injection

SECONDARY OUTCOMES:
Glabella line improvement rate at maximum frown confirmed with investigator's assessment (Phase II) | 8, 12 weeks after the injection
Glabellar line improvement rate at rest confirmed with investigator's assessment (Phase II) | 4, 8, 12 weeks after the injection
Glabellar line improvement rate at rest confirmed with subject's assessment (Phase II) | 4, 8, 12 weeks after the injection
Number of participants with treatment-related adverse events as assessed by CTCAE Version 5.0 (Phase II) | Up tp 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nowon Eulji Medical Center, Eulji University, Seoul, South Korea